CLINICAL TRIAL: NCT02557724
Title: Mobilization of Mesenchymal Stem Cells During Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Yuriy Gubenko, MD, Associate Professor, Department of Anesthesiology, Rutgers - NJMS, Rutgers, The State University of New Jersey
Other Study IDs: 20140000266
Record Dates: First submitted 2015-09-18; First posted 2015-09-23 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Liver Failure; Liver Neoplasm
MeSH Terms: conditions — Liver Failure; Liver Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- liver transplant patients: 5 blood samples at time points as described in protocol
  Interventions: Procedure: blood samples
- Liver resection patients: 3 blood samples at time points described in protocol
  Interventions: Procedure: blood samples

INTERVENTIONS:
Procedure: blood samples — liver transplant patients will have (5) 3cc blood samples drawn at specific time points.
  Groups: liver transplant patients
Procedure: blood samples — liver resection patients will have (3) 3cc. blood samples drawn at specific time points
  Groups: Liver resection patients

SUMMARY:
To study if the administration of corticoid hinder or enhance the mobilization of Mesenchymal Stem Cells (MSCs) in the peripheral blood during liver transplantation and whether this affects the outcome with respect to graft versus host response.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) are a known immune modulator with significant immunosuppressive effects. MSCs have emerged as a promising frontier in human clinical trials. MSCs have been shown to be non-immunogenic making them capable of transplantation across allogeneic barrier. These qualities make MSCs an ideal candidate to study if they are involved in reducing the rejection of the graft, in this case, liver transplant. If so, the information would be highly significant as it would lead to significant reduction in use of immunosuppressants with the replacement of MSCs. This will serve dual purposes: reduced clinical problems associated with pharmacological immunosuppression (discussed in the next paragraph); additional help in the protection of the transplanted liver by the MSCs.

The use of immunosuppressants in particular is vital in organ transplantation including liver transplant patients. However, their use is accompanied by numerous drawbacks such as reactivation of viral hepatitis, opportunistic infections and other complications. If MSCs can be used to decrease the use of immunosuppressive agents in liver transplant patients it can lead to a significant decrease in morbidity and mortality as a consequence of liver transplantation.

Hepatic macrophages, ie Kupffer cells, have a known function of recruiting monocytes into the liver. They have been shown to have a proinflammatory effect by attracting monocytes into the liver. They also interact with hepatic stellate cells (HSCs) which have pro-fibrogenic functions. However, they have been shown to have anti-inflammatory effects as well, implicating a role in fibrosis regression. Hepatic macrophages are an interesting new target for therapeutic intervention and the effect of steroids on kupffer cells as well as their interaction with MSCs have not been fully explored.

Patient will be attached to standard American Society of Anesthesiologists (ASA) monitors including pulse oximetry, electrocardiogram, noninvasive blood pressure monitoring temperature and capnometry. Patients will be placed under general anesthesia with endotracheal intubation and controlled ventilation. As is customary for all liver surgeries, an arterial line will be inserted for blood pressure monitoring and for repeat blood samples. If indicated, a pulmonary artery catheter will be inserted.

Anesthesia will be maintained using a volatile agent. Paralysis will be provided using a non-depolarizing neuromuscular blocking agent of the anesthesiologist's choice.

As is standard practice hourly blood samples will be taken from the arterial line to analyze Protime(PT)/International Normalized Ratio (INR)/Complete Blood Count/electrolytes. Red Blood Cells, Fresh Frozen Plasma and platelets will be transfused as necessary.

As is customary liver transplant recipients will be given the customary dose of methylprednisolone for immune suppression in the anhepatic phase.

Intraoperatively, patients undergoing transplant will have three blood samples collected from the arterial line for study purposes. Each sample will contain 3cc of blood.

The time points for blood samples are as follows:

* Immediately after arterial line placement as a baseline
* In the anhepatic stage prior to steroid injection
* Two hours after administration of steroids Post-operatively, two additional 3 mL blood samples will be taken by a member of the study team. The first will be on postoperative day 1 prior to the administration of immunosuppressive drugs and the second sample on postoperative day five. Thus for liver transplant patients a total of 15 milliliters (mL) of blood over a period of 5 days will be collected for the study.

The administration of immunosuppression drugs and or dosage will not be altered as a component of the research study.

A tissue sample of the liver donor organ will also be taken to culture MCSs (exempt informed consent).

Control group patients will undergo liver resection. They will not receive the dose of methylprednisolone. Intra-operatively blood samples will be collected at these time points:

* immediately after arterial line placement
* two hours after liver resection. Postoperatively two additional 3-mL blood samples will be taken. The first will be taken on postoperative day one and the second on postoperative day five or on the day of discharge whichever comes sooner. These samples will be collected by a study team member. A total of 12mL of blood over a period of 5 days will be collected from the liver resection patients for study purposes.

All blood samples will be immediately delivered to Dr. Rameswhar's lab, located in MSB, E579. The relative frequency of MSCs present in the blood of the two groups will be assessed by flow cytometry. The data will be presented as the percentage of MSCs/106 mononuclear cells. Statistical analyses will be performed to determine if there are differences between the two groups of subjects.

In addition to the above studies with the donor liver, we will also treat liver cells with glucocorticoids and then examine the liver for changes in aquaporin. The reason for this modification is to determine if aquaporin increases the ability to accumulate water. This additional study will not change the samples since only a small (<1mg) of tissue will be sufficient.

ELIGIBILITY:
Inclusion Criteria:

* • Patients 21-80 capable of providing informed consent

  * ASA rating between 1-4
  * Patients undergoing liver transplant or liver surgery for the first time.

Exclusion Criteria:

* • Patient less than 21 years of age

  * Patients unwilling to consent
  * If donor liver was obtained after cardiac death

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplant or liver resection
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
post operative liver injury | 0-7 post operative days
  . Primary endpoint is defined by postoperative liver injury assessed by peak serum value of aspartate aminotransferase (AST) or alanine aminotransferase (ALT).

SECONDARY OUTCOMES:
Total Bilirubin level | post operative day 7
  bilirubin greater than or equal to 10mg/dl on day 7
(INR) International Normalized Ratio | post operative day 7
  INR> or = to 1.6
(ALT) Alanine Aminotransferase | post operative day 7
  ALT> 2000 IU/L
(AST) Aspartate Aminotransferase | post operative day 7
  AST> 2000 IU/L

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Gubenko, MD, Principal Investigator — Rutrgers/SUNJ
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided